CLINICAL TRIAL: NCT02841514
Title: The Efficacy and Safety of Tooth Bleaching Procedure Using Y10 Whitening Toothpaste and RF Current
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: Brighttonix Medical Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CLD0043
Record Dates: First submitted 2016-07-18; First posted 2016-07-22 (Estimated); Last update posted 2019-07-10 (Actual); Status verified 2019-07

CONDITIONS: Tooth Bleaching

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- treatment group (Experimental): the operator will administer the Y10 whitening toothpaste in to the attachable mouthpiece and place it in the subject's mouth and turn on the device RF. After treating the patients for 30 minutes the operator will turn off the device and retrieve the mouthpiece from the mouth.
  Interventions: Device: The Y10 Tooth Whitening system including the Y10 toothpaste and the Y10 device
- placebo group (Placebo Comparator): the operator will administer an off the shelf regular toothpaste in to the attachable mouthpiece and place it in the subject's mouth. At this point the operator will switch on the device but the RF will not be activated. After 30 minutes the operator will turn off the device and retrieve the mouthpiece from the mouth.
  Interventions: Other: OTC toothpaste and an unoperated Y10 device

INTERVENTIONS:
Device: The Y10 Tooth Whitening system including the Y10 toothpaste and the Y10 device
  Arms: treatment group
Other: OTC toothpaste and an unoperated Y10 device
  Arms: placebo group

SUMMARY:
Study title: The Efficacy and Safety of tooth bleaching procedure using Y10 Whitening toothpaste and RF current

The Device: The Brighttonix Y10 Tooth Whitening system is indicated for use in painless non-invasive tooth whitening treatments.

Design: Single center, randomized, controlled, double blind, two-arm, prospective clinical study.

Follow up visits at 7 days (phone visit), 12 weeks and 26 weeks.

DETAILED DESCRIPTION:
Purpose: To assess the efficacy and the safety of tooth bleaching procedure using Y10 Whitening toothpaste and RF current (Y10 Device), versus placebo (no RF current and off- the -shelf non bleaching toothpaste) in healthy patients seeking tooth bleaching.

No. of Subjects/Sites: A total of 60 patients at Hadassah Medical Center will be randomized, 30 patients for the test arm, and 30 patients for the placebo arm.

A 40% to 60% male (or female) ratio will be maintained.

Target teeth: At least 4 teeth between teeth 13-23 (Upper front teeth) according to the international teeth numbering system.

Upper and lower teeth will be treated with the same treatment arm as described.

Endpoints:

Primary endpoint:

• At the end of the treatment (V3), compared to prior of treatment, the mean shade change will be at least two shades (Vita Bleachguide 3D Master, Vita P/N: B361) as measured at the middle one-third area of the labial surface of the selected target teeth.

Secondary endpoints:

* Compared to prior of treatment, the mean shade change at 3 and 6 months will be at least one shade (Vita Bleachguide 3D Master, Vita P/N: B361) as measured at the middle one-third area of the labial surface of the selected target teeth.
* Compared to prior of treatment, color change evaluates with a spectrophotometer (VITA Easyshade Advance 4; VITA Zahnfabrik, Bad Sackingen, Germany), before and after treatment, at 3 and 6 months will be at least one shade. (Device with a high reliability, over 96%, Kim-Pusateri Et al. Reliability and accuracy of four dental shade-matching devices. Journal of Prosthetic Dentistry United States 2009;101(March (3)):193-9.)
* Compared to prior of treatment, the mean shade change for the lower teeth numbers 43-33 after treatment, 3 and 6 months will be at least one shade.
* Lesion in the gingiva of the upper and lower teeth (+/- in each of the teeth numbers 33-43, 13-23 after treatment and 3 months.
* Compared to prior of treatment - teeth sensitivity to cold and touch stimulation - target teeth - VAS scale after treatment, 3 and 6 months. For the VAS, the participants will place a line perpendicular to a 10-mm-long line with zero at one end indicating ''no TS'' and the other end indicating ''unbearable TS.''
* Patient oral questionnaire - post treatment, 7 days, 3 months, 6 months (See below).
* Patient Reported Outcomes: (Scale 0-4). OHIP14-aesthetics questions for patients that received dental bleaching - (see below) - before treatment and in 3 months.
* Periodontal parameters at baseline, 3 and 6 months: plaque index, sulcular bleeding index, pocket depth - all at the target teeth. (See below details).

Inclusion criteria:

1. Signed and dated Informed Consent Form.
2. Normal and controlled general health.
3. Male or female patients aged between 18-60 years old.
4. Availability for the 37 weeks duration of the study.
5. The patient has at least 4 natural teeth with no buccal restoration in the upper front area of the jaw (teeth 13-23), at least 2 of them with VITA shade >15, in accordance with VITA Bleachedguide 3D-MASTER (P/N: B361, VITA Zahnfabrik H Rauter GmbH & Co. KG, D-79713 Bad Sackingen, Germany).
6. Females of childbearing potential must be non-pregnant or non-lactating during the course of the study

Exclusion criteria:

1. Underwent a teeth bleaching procedure in the last 3 years.
2. Pockets of >5 mm with BOP in the target area.
3. Heavy smokers - > 10 cigarettes per day.
4. Tetracycline staining of target teeth.
5. Presence of oral local mechanical factors that could (in the opinion of the Investigator) influence the outcome of the study.
6. Presence of dental restorations in more than 2 teeth in the target area.
7. Uncontrolled periodontitis or sever gingival inflammation
8. Scheduled or simultaneous periodontal treatment.
9. Presence of orthodontic appliances, or any removable appliances.
10. Presence of soft or hard tissue tumours of the oral cavity.
11. Presence of any of the following oral conditions: major recurrent aphthous ulcers, stomatitis, abscesses and related oral pathologies.
12. The presence of any medical or psychiatric condition or any other condition that, in the opinion of the Investigator, could affect the successful participation of the patient in the study.
13. Subject participates in any other clinical study 30 days prior to the start of the study and throughout the study duration.
14. Implanted pacemaker or internal defibrillator, or any other active electrical implant anywhere in the body
15. Medical conditions of bleeding disorders, leukaemia, cirrhosis, vascular disease, sarcoidosis, active hepatitis, HIV.

ELIGIBILITY:
Inclusion Criteria:

1. Signed and dated Informed Consent Form.
2. Normal and controlled general health.
3. Male or female patients aged between 18-60 years old.
4. Availability for the 37 weeks duration of the study.
5. The patient has at least 4 natural teeth with no buccal restoration in the upper front area of the jaw (teeth 13-23), at least 2 of them with VITA shade >15, in accordance with VITA Bleachedguide 3D-MASTER (P/N: B361, VITA Zahnfabrik H Rauter GmbH & Co. KG, D-79713 Bad Sackingen, Germany).
6. Females of childbearing potential must be non-pregnant or non-lactating during the course of the study

Exclusion Criteria:

1. Underwent a teeth bleaching procedure in the last 3 years.
2. Pockets of >5 mm with BOP in the target area.
3. Heavy smokers - > 10 cigarettes per day.
4. Tetracycline staining of target teeth.
5. Presence of oral local mechanical factors that could (in the opinion of the Investigator) influence the outcome of the study.
6. Presence of dental restorations in more than 2 teeth in the target area.
7. Uncontrolled periodontitis or sever gingival inflammation
8. Scheduled or simultaneous periodontal treatment.
9. Presence of orthodontic appliances, or any removable appliances.
10. Presence of soft or hard tissue tumours of the oral cavity.
11. Presence of any of the following oral conditions: major recurrent aphthous ulcers, stomatitis, abscesses and related oral pathologies.
12. The presence of any medical or psychiatric condition or any other condition that, in the opinion of the Investigator, could affect the successful participation of the patient in the study.
13. Subject participates in any other clinical study 30 days prior to the start of the study and throughout the study duration.
14. Implanted pacemaker or internal defibrillator, or any other active electrical implant anywhere in the body
15. Medical conditions of bleeding disorders, leukaemia, cirrhosis, vascular disease, sarcoidosis, active hepatitis, HIV.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2016-09; Primary Completion 2017-04 (Estimated)

PRIMARY OUTCOMES:
At the end of the treatment (V3), compared to prior of treatment, the mean shade change will be at least two shades (Vita Bleachguide) as measured at the middle one-third area of the labial surface of the selected target teeth. | 26 weeks

SECONDARY OUTCOMES:
Compared to prior of treatment, the mean shade change at 3 and 6 months will be at least one shade (Vita Bleachguide) as measured at the middle one-third area of the labial surface of the selected target teeth. | up to 26 weeks
Compared to prior of treatment, color change evaluates with a spectrophotometer (VITA Easyshade) before and after treatment, at 3 and 6 months will be at least one shade. | up to 26 weeks
Compared to prior of treatment, the mean shade change for the lower teeth numbers 43-33 after treatment, 3 and 6 months will be at least one shade. | up to 26 weeks
Lesion in the gingiva of the upper and lower teeth (+/- in each of the teeth numbers 33-43, 13-23 after treatment and 3 months. | 12 weeks
Compared to prior of treatment - teeth sensitivity to cold and touch stimulation - target teeth - VAS scale after treatment, 3 and 6 months. | up to 26 weeks
Patient oral questionnaire - post treatment, 7 days, 3 months, 6 months. | up to 26 weeks
Patient Reported Outcomes: (Scale 0-4). OHIP14-aesthetics questions for patients that received dental bleaching - (see below) - before treatment and in 3 months. | 12 weeks
Periodontal parameters at baseline, 3 and 6 months: plaque index - all at the target teeth. | up to 26 weeks
Periodontal parameters at baseline, 3 and 6 months: sulcular bleeding index- all at the target teeth. | up to 26 weeks
Periodontal parameters at baseline, 3 and 6 months: pocket depth - all at the target teeth. | up to 26 weeks